CLINICAL TRIAL: NCT01501253
Title: Evaluate the Efficacy and Safety of a Fixed Dose Combination of S-Amlodipine and Telmisartan(CKD-828) vs. S-Amlodipine Monotherapy in Hypertensive Patients Inadequately Controlled by S-Amlodipine Monotherapy.
Brief Title: CKD-828 S-Amlodipine Non-Responder Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130HT11A
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: CKD-828; Hypertension; Primary Hypertension; S-Amlodipine; Telmisartan; Non-Responder
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — levamlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CKD-828 2.5/40mg (Experimental): CKD-828 2.5/40mg
  Interventions: Drug: CKD-828 2.5/40mg
- CKD-828 2.5/80mg (Experimental): CKD-828 2.5/80mg
  Interventions: Drug: CKD-828 2.5/80mg
- S-Amlodipine 2.5mg (Active Comparator): S-Amlodipine 2.5mg
  Interventions: Drug: S-Amlodipine 2.5mg

INTERVENTIONS:
Drug: CKD-828 2.5/40mg — fixed dose combination of S-Amlodipine 2.5mg and Telmisartan 40mg
  Arms: CKD-828 2.5/40mg
Drug: CKD-828 2.5/80mg — Fixed dose combination of S-Amlodipine 2.5 and Telmisartan 80mg
  Arms: CKD-828 2.5/80mg
Drug: S-Amlodipine 2.5mg — S-Amlodipine 2.5mg monotherapy
  Other Names: Anydipine S tab.
  Arms: S-Amlodipine 2.5mg

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of two dose combination of S-Amlodipine/Telmisartan (2.5/40mg amd 2.5/80mg) compared with S-Amlodipine monotherapy (2.5mg) in hypertensive patients inadequately controlled by S-Amlodipine monotherapy.

DETAILED DESCRIPTION:
* In patients with essential hypertension inadequately controlled by S-Amlodipine monotherapy to evaluate the efficacy and safety of two dose combination of S-Amlodipine/Telmisartan (2.5/40mg amd 2.5/80mg) compared with S-Amlodipine monotherapy (2.5mg)during 8weeks.
* Included S-Amlodipine run-in period(during 4 weeks_single blind) and Treatment period(during 8 weeks_double blind).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* diagnosis of essential hypertension and blood pressure not adequately controlled (inadequate control defined as seated diastolic blood pressure(DBP)≥ 90mmHg if on existing amtihypertensive treatment of seated DBP≥100mmHg if treatment naive)
* failure to respond to four weeks treatment with S-Amlodipine 2.5mg(failure to respond defined as seated DBP ≥ 90mmHg)
* willing and able to provide written informed consent

Exclusion Criteria:

* mean seated DBP ≥ 120mmHg and/or mean seated SBP ≥ 200mmHg during run-in treatment or mean seated DBP ≥ 120mmHg and/or mean seated SBP ≥ 180mmHg at the randomization visit
* known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* has severe heart disease(Heart failure NYHA functional class 3, 4), unstable angina or myocardial infarction, arrhythmia within the past three months
* has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabetes Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c) > 8%
* known severe or malignant retinopathy
* hepatic or renal dysfunction as defined by the following laboratory parameters: AST/ALT > UNL X 2, serum creatinine > UNL X 1.5
* acute or chronic inflammatory status need to treatment
* need to additional antihypertensive drugs during the study
* need to concomitant medications known to affect blood pressure during the study
* history of angioedema related to ACE inhibitors or Angiotensin II Receptor Blockers
* known hypersensitivity related to either study drug
* history of drug or alcohol dependency within 6 months
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, gastric ulcers need to treatment, gastrointestinal/rectal bleeding, impaired pancreatic function such as pancreatitis, obstructions of the urinary tract or difficulty in voiding
* administration of other study drugs within 30 days prior to randomization
* premenopausal women(last menstruation < 1year) not using adequate contraception, pregnant or breast-feeding
* history of malignancy including leukemia and lymphoma within the past 5 years
* in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 8 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 4 weeks of treatment
Mean Sitting Systolic Blood Pressure (MSSBP) | After 4 weeks and 8 weeks of treatment
Control Rate | After 8 weeks of treatment
  SBP<140mmHg, DBP<90mmHg
Response Rate | After 8 weeks of treatment
  Reduction of SBP≥20mmHg, DBP≥10mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Joong Yoon, Ph.D, Principal Investigator — Seoul St. Mary's hospital, The catholic university of Korea
Locations (1):
- Seoul St. Mary's hospital, The catholic university of Korea, Seoul, South Korea